CLINICAL TRIAL: NCT06135675
Title: A Phase 1b/2a Study to Evaluate the Safety, Tolerability, PK Profile and Preliminary Efficacy of Multiple Doses of TNP-2092 Capsules in Liver Cirrhosis Patients With Hyperammonemia
Brief Title: PK Profile and Preliminary Efficacy of TNP-2092 Capsules in Liver Cirrhosis Patients With Hyperammonemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TenNor Therapeutics (Suzhou) Limited (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TNP-2092-06
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Hyperammonemia
MeSH Terms: conditions — Hyperammonemia | interventions — TNP-2092

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TNP-2092 capsules 100mg Twice daily(BID) (Experimental): Subjects received TNP-2092 capsules orally twice daily at the dose of 100 mg in the fed state for consecutive 14 days and received the last dose in the fed state on the morning of Day 15.
  Interventions: Drug: TNP-2092 capsules
- TNP-2092 capsules 300mg BID (Experimental): Subjects received TNP-2092 capsules orally twice daily at the dose of 300 mg in the fed state for consecutive 14 days and received the last dose in the fed state on the morning of Day 15.
  Interventions: Drug: TNP-2092 capsules
- TNP-2092 capsules 600mg BID (Experimental): Subjects received TNP-2092 capsules orally twice daily at the dose of 600 mg in the fed state for consecutive 14 days and received the last dose in the fed state on the morning of Day 15.
  Interventions: Drug: TNP-2092 capsules
- Placebo (Placebo Comparator): Subjects received TNP-2092 placebo capsules orally twice daily in the fed state for consecutive 14 days and received the last dose in the fed state on the morning of Day 15.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TNP-2092 capsules — Administration orally.
  Other Names: Rifaquizinone capsules
  Arms: TNP-2092 capsules 100mg Twice daily(BID); TNP-2092 capsules 300mg BID; TNP-2092 capsules 600mg BID
Drug: Placebo — Administration orally.
  Other Names: TNP-2092 placebo capsules
  Arms: Placebo

SUMMARY:
The aim of this study was to evaluate the safety, tolerability, and pharmacokinetic characteristics of TNP-2092 Capsules in liver cirrhosis patients with hyperammonemia; and to preliminarily observe the effects of the study drug on blood ammonia and hepatic encephalopathy related clinical symptoms and signs, neuropsychological indicators, and quality of life in liver cirrhosis patients with hyperammonemia.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the safety, tolerability, and pharmacokinetic characteristics of TNP-2092 Capsules in liver cirrhosis patients with hyperammonemia; and to preliminarily observe the effects of the study drug on blood ammonia and hepatic encephalopathy related clinical symptoms and signs, neuropsychological indicators, and quality of life in liver cirrhosis patients with hyperammonemia.

A total of 3 dose groups will be set up, i.e., 100 mg BID, 300 mg BID and 600 mg BID groups. Drugs will be orally administered 30 min after breakfast and dinner for 14 consecutive days, and last dose will be administered 30 min after breakfast on the morning of D15. Each dose group will include a study drug TNP-2092 capsule arm and a placebo control arm. Subjects will exit upon completion of the safety and tolerability evaluation on D17.

Twelve liver cirrhosis patients with hyperammonemia are planned to be enrolled in each dose group. The 12 patients will be assigned in a ratio of 2:1 to the TNP-2092 capsule arm and the placebo arm, with 8 patients receiving TNP-2092 Capsules and 4 receiving placebos.

Enrollment for the second dose group may start only after the previous dose group has fully completed the treatment period and passed the safety and tolerability evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 (inclusive) years of age, male or female.
* Clinically diagnosed with liver cirrhosis.
* Fasting venous blood ammonia above upper limit of normal (ULN).
* Organ functions must meet the following criteria:
* Peripheral blood: absolute neutrophil count ≥ 0.5*109/L, platelet ≥20*109/L, hemoglobin ≥ 8 g/dL.
* Liver: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × ULN; serum total bilirubin (TBL) ≤ 5 × ULN.
* Kidney: creatinine clearance ≥ 60 mL/min.
* No malabsorption or other gastrointestinal disorders that affect drug absorption.
* Weight ≥ 45 kg and body mass index [BMI = weight (kg)/height 2 (m2) ] between 18 and 34 (inclusive) kg/m2.
* Subjects (including their partners) will have no pregnancy plan and voluntarily take effective contraceptive measures within 6 months after drug withdrawal. Refer to Appendix 9 for specific contraceptive measures.
* Subjects or their legal representatives sign the Informed Consent Form and fully understand the content, procedures, and potential adverse reactions prior to the initiation of the study.
* Able to complete the study per the requirements in the study protocol.

Exclusion Criteria:

* Subjects who are allergic to rifamycin or quinolone antibacterial agents or those with an allergic constitution.
* Pregnant or lactating women, or women of childbearing age with a positive pregnancy test from the screening period to initiation of the study treatment.
* Subjects with serious nervous or mental disorders.
* Subjects with Child-Pugh class C liver cirrhosis.
* Subjects with Grade 2 or above hepatic encephalopathy.
* Subjects who have been diagnosed with Clostridium difficile-induced pseudomembranous enteritis within 3 months.
* Subjects who have had systemic infection or gastrointestinal bleeding within 7 days prior to screening.
* Subjects with clinically significant abnormal clinical laboratory tests or other clinical findings indicative of clinically significant disorders that, in the opinion of the investigator, make them not eligible for this clinical study.
* Subjects who have used sedatives, probiotics, cathartics or antibacterial agents within 7 days prior to screening.
* Subjects who have used other study drugs or participated in other drug clinical trials within 1 month prior to screening.
* Subjects need to use the following concomitant drugs during the study treatment period: cathartics and drugs for ammonia reduction listed in 5.2.1 in the Guidelines on the Management of Hepatic Encephalopathy in Liver Cirrhosis 2018 (e.g., lactulose, lactitol, L-ornithine L-aspartate(LOLA), rifaximin, other antibacterial agents, etc.) ; HIV protease inhibitors (e.g., ritonavir boosted or non-boosted saquinavir, atazanavir, darunavir, fosamprenavir, tipranavir, etc.) ; praziquantel; halothane; class IA and III antiarrhythmics (disopyramide, procainamide, quinidine, amiodarone, dofetilide, dronedarone, ibutilide, sotalol, etc.) ; strong inhibitors and inducers of liver metabolic enzymes;
* Positive HIV antigen/antibody screen; positive Treponema pallidum antibody screen requires the investigator's judgment with the consideration of Rapid plasma regain（RPR） results.
* Positive urine drug screen or history of drug abuse within the past 5 years.
* Positive alcohol breath test.
* Acute diseases or concomitant medications from screening to study medication.
* Other circumstances deemed by the investigator to be unsuitable for enrollment in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TNP-2092 Capsules 100mg Twice Daily(BID); TNP-2092 Capsules 300mg BID; TNP-2092 Capsules 600mg BID: TNP-2092 capsules: TNP-2092 capsules will be orally administered 30 min after breakfast and dinner for 14 consecutive days, and last dose will be administered 30 min after breakfast on the morning of D15.
- TNP-2092 Capsules Placebo: TNP-2092 capsules Placebo: TNP-2092 capsules Placebo will be orally administered 30 min after breakfast and dinner for 14 consecutive days, and last dose will be administered 30 min after breakfast on the morning of D15.
Period: Overall Study
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID | TNP-2092 Capsules Placebo
Started | 8 | 8 | 8 | 12
Completed | 7 | 8 | 8 | 11
Not Completed | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID | TNP-2092 Capsules Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 12 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (7.19) | 50.4 (5.71) | 51.9 (7.97) | 52.3 (10.15) | 51.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 4 | 8
  Male | 8 | 7 | 5 | 8 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 8 | 8 | 12 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Fasting Venous Blood Ammonia Concentration [Mean (Standard Deviation); unit: μmol/L] — Fasting venous blood ammonia concentration before first dosing.
  μmol/L | 90.1 (27.1) | 80.3 (19.5) | 78.8 (17.3) | 115.8 (39.1) | 94.0 (32.0)

OUTCOME MEASURES:

1. Primary Outcome: Safety of TNP-2092 by Assessment of the Number of Participants With Adverse Events (AEs)
Description: To investigate the safety and tolerability of TNP-2092 by assessment of the number of participants with AEs following administration of TNP-2092 capsules. An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 17 days after the first dosing.
Population: All subjects who have received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 12
participants | 6 | 6 | 7 | 8

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of TNP-2092 Capsules in Liver Cirrhosis Patients With Hyperammonemia on Day 1.
Description: Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma PK parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Time Frame: Day 1: 30-60 min prior to the first dose, and 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h and 12 h post-dose
Population: All subjects who have been randomized into groups, have received at least one dose of study drug, and have at least one evaluable pharmacokinetic parameter.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 8 | 8 | 8
ng/ml | 90.4 (42.9) | 140 (120) | 415 (294)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Administration to the Time of the Last Measurable Plasma Concentration (AUC0-last) on Day 1.
Description: as for outcome 2
Time Frame: Day 1: 30-60 min prior to the first dose, and 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h and 12 h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 8 | 8 | 8
h*ng/ml | 309 (178) | 524 (537) | 1610 (1200)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Administration Extrapolated to Infinity (AUC0-∞) on Day 15
Description: as for outcome 2
Time Frame: Day 15: 30-60 min prior to the first dose, and 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h, 24 h and 36 h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 7 | 8 | 8
h*ng/ml | 396 (257) | 756 (570) | 2680 (1790)

5. Primary Outcome: Time to Reach the Maximum Observed Plasma Concentration (Tmax) on Day 1
Description: as for outcome 2
Time Frame: Day 1: 30-60 min prior to the first dose, and 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h and 12 h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 8 | 8 | 8
h | 4.75 (0.46) | 5.13 (0.36) | 5.13 (0.35)

6. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of TNP-2092 Capsules in Liver Cirrhosis Patients With Hyperammonemia on Day 15.
Description: as for outcome 2
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 7 | 8 | 8
ng/ml | 60.8 (28.5) | 164 (118) | 543 (420)

7. Primary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Administration to the Time of the Last Measurable Plasma Concentration (AUC0-last) on Day 15.
Description: as for outcome 2
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 7 | 8 | 8
h*ng/ml | 380 (247) | 739 (555) | 2610 (1730)

8. Primary Outcome: Time to Reach the Maximum Observed Plasma Concentration (Tmax) Day 15
Description: as for outcome 2
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 7 | 8 | 8
h | 4.43 (0.78) | 4.75 (0.46) | 4.50 (1.85)

9. Primary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Administration Extrapolated to Infinity (AUC0-∞) Day 1
Description: as for outcome 2
Time Frame: Day 1: 30-60 min prior to the first dose, and 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h and 12 h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 8 | 8 | 8
h*ng/ml | 332 (188) | 561 (565) | 1790 (1210)

10. Primary Outcome: Half Life (t1/2) of TNP-2092 Capsules on Day 1
Description: as for outcome 2
Time Frame: Day 1: 30-60 min prior to the first dose, and 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h and 12 h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 8 | 8 | 8
h | 2.52 (0.63) | 2.23 (0.81) | 2.99 (2.29)

11. Primary Outcome: Half Life (t1/2) of TNP-2092 Capsules on Day 15
Description: as for outcome 2
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 8 | 8 | 8
h | 8.17 (1.84) | 6.92 (2.63) | 7.93 (1.09)

12. Primary Outcome: Area Under the Plasma Concentration-time Curve Within a Dosing Interval (AUC0-tau) on Day 1
Description: as for outcome 2
Time Frame: Day 1: 30-60 min prior to the first dose, and 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h and 12 h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 309 (179) | 525 (538) | 1610 (1200)

13. Primary Outcome: Area Under the Plasma Concentration-time Curve Within a Dosing Interval (AUC0-tau) on Day 15
Description: as for outcome 2
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 303 (187) | 646 (466) | 2230 (1480)

14. Primary Outcome: Accumulation Index Rac(Cmax) of TNP-2092 Capsules in Liver Cirrhosis Patients With Hyperammonemia
Description: Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma PK parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
  Rac (Cmax) was calculated from the ratio of Cmax (Day 15) to Cmax (Day 1)
Time Frame: Day 1: 30-60 min prior to first dose, and 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, and 12 h post-dose (prior to next dose). Day 15: 30-60 min pre-dose, and 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h, 24 h and 36 h post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 8 | 8 | 8
ratio | 0.74 (0.22) | 1.23 (0.49) | 1.26 (0.42)

15. Primary Outcome: Accumulation Index Rac(AUC) of TNP-2092 Capsules in Liver Cirrhosis Patients With Hyperammonemia
Description: Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma PK parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
  Rac (AUC) was calculated from the ratio of AUC0-tau (Day 15) to AUC0-tau(Day 1).
Time Frame: as for outcome 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID
Number analyzed (Participants) | 8 | 8 | 8
ratio | 1.09 (0.40) | 1.38 (0.39) | 1.47 (0.55)

16. Secondary Outcome: Changes in the Fasting Venous Blood Ammonia Concentration From Baseline (Mean Pre-treatment Measured)
Description: The changes in the fasting venous blood ammonia concentration from baseline will be compared with the placebo to evaluate the preliminary efficacy of TNP-2092 Capsules in liver cirrhosis patients with hyperammonemia.
Time Frame: Baseline and Day 15
Population: All the subjects who were randomized into groups
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 12
μmol/L | 5.7 (17.50) | -2.1 (22.49) | -14.1 (18.12) | 0.5 (45.29)

17. Secondary Outcome: Proportion of Participants With Positive Result of Number Connection Test A (NCT-A)
Description: Evaluation of NCT-A is based on the time required to complete the test. The results will be positive according to following criteria: 1) the time is over 34.3 seconds while the age is less than 35 years; 2) the time is over 45.7 seconds while the age is between 35 to 44 years; 3) the time is over 52.8 seconds while age is between 45 to 54 years; 4) the time is over 61.9 seconds while the age is between 55 to 64 years.
  The positive result means a worse outcome.
Time Frame: Baseline, Day 7 and Day 15
Population: All the subjects who were randomized into groups
Measure: Count of Participants; unit: Participants
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 12
Participants
  Baseline | 6 | 6 | 8 | 12
  Day 7 | 7 | 6 | 8 | 12
  Day 15 | 5 | 7 | 8 | 11

18. Secondary Outcome: Proportion of Participants With Positive Result of Digital Symbol Test (DST)
Description: Evaluation of Digital symbol test (DST) is based on the score gained within 90 seconds, and the results are positive according to following criteria: 1) the score is less than 40.5 while the age is less than 35 years; 2) the score is less than 35.0 while the age is between 35 to 44 years; 3) the score is less than 28.5 while the age is between 45 to 54 years; 4) the score is less than 26.0 while the age is between 55 to 64 years.
  The positive result means a worse outcome.
Time Frame: Baseline, Day 7 and Day 15
Population: All the subjects who were randomized into groups
Measure: Count of Participants; unit: Participants
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 12
Participants
  Baseline | 4 | 2 | 3 | 7
  Day 7 | 4 | 2 | 3 | 8
  Day 15 | 0 | 1 | 3 | 7

19. Secondary Outcome: Changes in the Total Scores of Quality of Life (QOL) From Baseline
Description: Changes in the total scores of QOL from baseline will be compared with the placebo to evaluate the preliminary efficacy of TNP-2092 Capsules in liver cirrhosis patients with hyperammonemia. The range of QOL scores is 30 ~ 150. Patients with lower scores means a better outcome.
Time Frame: Baseline, Day 7 and Day 15
Population: All the subjects who were randomized into groups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 12
score on a scale
  Day 7 | -6.1 (5.64) | 6.4 (15.80) | 3.1 (13.91) | 0.5 (9.21)
  Day 15 | -3.0 (4.73) | 7.1 (15.82) | 4.6 (5.63) | -1.4 (15.88)

20. Secondary Outcome: Proportion of Participants Whose Asterixis is Elicited
Description: Asterixis is a physical exam finding that can be elicited by asking the participant to extend the arms, flex the wrists, and spread the fingers wide. Clinically, asterixis produces flapping tremors. In a flapping tremor, an participant will flap their wrists like a bird flapping its wings.
  Asterixis elicited means a worse outcome.
Time Frame: Baseline, Day 7 and Day 15
Population: All the subjects who were randomized into groups
Measure: Count of Participants; unit: Participants
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 12
Participants
  Whether asterixis is elicited at Baseline: Yes | 0 | 0 | 0 | 0
  Whether asterixis is elicited at Baseline: No | 8 | 8 | 8 | 12
  Whether asterixis is elicited on Day 7: Yes | 0 | 0 | 0 | 0
  Whether asterixis is elicited on Day 7: No | 8 | 8 | 8 | 12
  Whether asterixis is elicited on Day 15: Yes | 0 | 0 | 0 | 0
  Whether asterixis is elicited on Day 15: No | 8 | 8 | 8 | 12

21. Secondary Outcome: Clinical Grade of Hepatic Encephalopathy
Description: Grade 0 of HE (without HE) is nomal, Grade 0 of HE (MHE) is alterations of brain function in neuropsychological or neurophysiological measures without clinical signs of HE, Grade 1 of HE is mild lack of awareness, Grade 2 of HE is lethargic, Grade 3 of HE is somnolent, and Grade 4 of HE is coma.
  Higher score means worse outcome.
Time Frame: Baseline, Day 7 and Day 15
Population: All the subjects who were randomized into groups
Measure: Count of Participants; unit: Participants
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 12
Participants
  Baseline: Grade 0 of HE (without HE) | 2 | 2 | 0 | 0
  Baseline: Grade 0 of HE (MHE) | 6 | 6 | 8 | 12
  Baseline: Grade 1 of HE | 0 | 0 | 0 | 0
  Baseline: Grade 2 of HE | 0 | 0 | 0 | 0
  Baseline: Grade 3 of HE | 0 | 0 | 0 | 0
  Baseline: Grade 4 of HE | 0 | 0 | 0 | 0
  Day 7: Grade 0 of HE (without HE) | 1 | 1 | 0 | 0
  Day 7: Grade 0 of HE (MHE) | 7 | 7 | 8 | 12
  Day 7: Grade 1 of HE | 0 | 0 | 0 | 0
  Day 7: Grade 2 of HE | 0 | 0 | 0 | 0
  Day 7: Grade 3 of HE | 0 | 0 | 0 | 0
  Day 7: Grade 4 of HE | 0 | 0 | 0 | 0
  Day 15: Grade 0 of HE (without HE) | 1 | 1 | 0 | 0
  Day 15: Grade 0 of HE (MHE) | 7 | 7 | 8 | 12
  Day 15: Grade 1 of HE | 0 | 0 | 0 | 0
  Day 15: Grade 2 of HE | 0 | 0 | 0 | 0
  Day 15: Grade 3 of HE | 0 | 0 | 0 | 0
  Day 15: Grade 4 of HE | 0 | 0 | 0 | 0

22. Secondary Outcome: Areas Under the Blood Ammonia Concentration-time Curve
Description: Plasma concentrations of Blood Ammonia were measured by a specific and validated assay. Changes in the Fasting Venous Blood Ammonia Concentration From Baseline were used to measure AUC.
Time Frame: Baseline to Day 15
Population: All the subjects who were randomized into groups
Measure: Mean (Standard Deviation); unit: h*μmol/L
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 12
h*μmol/L
  Day 1 | 481.6 (564.5) | 480.2 (607.9) | 225.0 (544.1) | 85.5 (999.3)
  Day 1-Day 15 | -1716.7 (5778.5) | -3205.4 (8311.8) | -5805.6 (6080.5) | -5476.3 (12816.5)

ADVERSE EVENTS:
Time Frame: 17 days after the first dose
Arm/Group | TNP-2092 Capsules 100mg Twice Daily(BID) | TNP-2092 Capsules 300mg BID | TNP-2092 Capsules 600mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 1/12
Other Adverse Events (participants affected / at risk) | 6/8 | 6/8 | 7/8 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNP-2092 Capsules 100mg Twice Daily(BID) (N=8) | TNP-2092 Capsules 300mg BID (N=8) | TNP-2092 Capsules 600mg BID (N=8) | Placebo (N=12)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNP-2092 Capsules 100mg Twice Daily(BID) (N=8) | TNP-2092 Capsules 300mg BID (N=8) | TNP-2092 Capsules 600mg BID (N=8) | Placebo (N=12)
neutrophil count decreased (Investigations) | 2 (4) | 4 (6) | 6 (7) | 6 (7)
white blood cell count decreased (Investigations) | 2 (2) | 2 (3) | 6 (7) | 4 (4)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (4) | 4 (5) | 2 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 1 (2) | 2 (2)
Platelet count decreased (Investigations) | 3 (4) | 1 (5) | 0 (0) | 5 (5)
Lipase increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood fibrinogen decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT06135675/Prot_SAP_000.pdf